CLINICAL TRIAL: NCT03517228
Title: Pilot Trial of the Robotic Uterine Manipulator
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Enrollment incomplete
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: Northwell Health (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 18-173
Record Dates: First submitted 2018-04-24; First posted 2018-05-07 (Actual); Results first posted 2024-08-07 (Actual); Last update posted 2024-09-04 (Actual); Status verified 2024-08

CONDITIONS: Gynecologic Surgery
Keywords: Robotic Uterine Manipulator; 18-173

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- total laparoscopic or robotic-assisted hysterectomy (Experimental): All patients who are consented for a total laparoscopic or robotic-assisted hysterectomy will be eligible for the trial, unless the surgeon does not plan to use a uterine manipulator.
  Interventions: Device: BAUM device

INTERVENTIONS:
Device: BAUM device — The robotic manipulator will be placed at the start of each case. The manipulator will be cleaned and sanitized using the same process as other reusable OR devices. Feasibility will be determined by the rate of successful robotic manipulator docking and if the manipulation of the uterus was successful for the duration of the procedure. The V-Care is an FDA approved uterine manipulator which will attach to the investigational BAUM. Placement of a BAUM will be noted on the operative note.

SUMMARY:
The purpose of this study is to test a robotic uterine manipulator system called the Barakat Automated Uterine Manipulator (BAUM), which will assist the surgeon in moving and positioning the uterus during a hysterectomy. This new device will allow the surgeon to control the movements of the robotic arm directly instead of giving verbal instructions to a staff member. The BAUM has never been used during surgeries before this trial. Overall, the study goal is to determine whether the use of this robotic uterine manipulator system can be safely used in the operating room while improving surgeon control during the procedure.

ELIGIBILITY:
Inclusion Criteria:

* Female participant must be scheduled for a total laparoscopic or robotic-assisted hysterectomy for a gynecologic condition
* Female participants must be 18 years of age or older

Exclusion Criteria:

* Female participant is not eligible if the surgeon does not plan to use a uterine manipulator

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — gynecologic surgery
Enrollment: 28 (Actual)
Dates: Start 2018-04-24 (Actual); Primary Completion 2023-12-12 (Actual); Study Completion 2023-12-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mario Leitao, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (7):
- United States (7):
  - Memorial Sloan Kettering Basking Ridge (Consent only), Basking Ridge, New Jersey
  - Memorial Sloan Kettering Monmouth (Consent only), Middletown, New Jersey
  - Memorial Sloan Kettering Bergen (Consent only), Montvale, New Jersey
  - Memorial Sloan Kettering Commack (Consent only), Commack, New York
  - Memorial Sloan Kettering Westchester (Consent only), Harrison, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Memorial Sloan Kettering Nassau (Consent only), Uniondale, New York

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/mskcc/html/44.cfm

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Total Laparoscopic or Robotic-assisted Hysterectomy
Started | 28
Completed | 18
Not Completed | 10
Not completed — Withdrawal by Subject | 2
Not completed — Hard drive issues, abandoned prior to surgery | 2
Not completed — Anatomy issue - abandoned prior to surgery | 1
Not completed — Surgery was at MAIN, could not change location to JOSIE | 1
Not completed — Canceled due to device being updated | 1
Not completed — No V Cares in stock | 1
Not completed — Service issue, use of device cancelled prior to surgery | 2

BASELINE CHARACTERISTICS:
Arm/Group | Total Laparoscopic or Robotic-assisted Hysterectomy
Number analyzed (Participants) | 28
Age, Continuous [Median (Full Range); unit: years] | 57 [38 to 75]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3
  Not Hispanic or Latino | 24
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 24
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 28

OUTCOME MEASURES:

1. Primary Outcome: the Number of Intraoperative Complications Attributed to the Robotic Manipulator.
Description: will be assessed by reporting all intraoperative complications during the surgery. Complications might include vaginal tear or uterine perforation.
Time Frame: 25- 35 days
Measure: Number; unit: # of intraoperative complications
Arm/Group | Total Laparoscopic or Robotic-assisted Hysterectomy
Number analyzed (Participants) | 28
# of intraoperative complications | 0

ADVERSE EVENTS:
Time Frame: Up to 35 days
Arm/Group | Total Laparoscopic or Robotic-assisted Hysterectomy
All-Cause Mortality (participants affected / at risk) | 3/28
Serious Adverse Events (participants affected / at risk) | 0/28
Other Adverse Events (participants affected / at risk) | 0/28

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-01-02): https://cdn.clinicaltrials.gov/large-docs/28/NCT03517228/Prot_SAP_000.pdf